CLINICAL TRIAL: NCT01689935
Title: A Pilot Clinical Trial to Reduce Side-Effects of Photodynamic Therapy for the Treatment of Moderate to Severe Acne
Brief Title: Reduced Side-Effects of Photodynamic Therapy for the Treatment of Moderate to Severe Acne (i-PDT)
Acronym: i-PDT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Richard Rox Anderson, MD, Professor, Harvard Medical School (Dermatology), Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-P-002352
Record Dates: First submitted 2011-10-05; First posted 2012-09-21 (Estimated); Last update posted 2025-02-20 (Actual); Status verified 2019-09

CONDITIONS: Acne Vulgaris
Keywords: Acne vulgaris; Photodynamic Therapy; Side-effects; Pain
MeSH Terms: conditions — Acne Vulgaris; Pain | interventions — Aminolevulinic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Control (No Intervention): No drug, no treatment
- ALA-PDT (Active Comparator): Drug- topical 20% Aminolevulinic acid - ALA followed by red light irradiation - conventional photodynamic therapy -PDT
  Interventions: Drug: 20 % Aminolevulinic Acid
- i-PDT (Experimental): Drug - topical 20% Aminolevulinic acid - followed by inhibitory light during incubation time, then red light for photodynamic therapy
  Interventions: Drug: 20 % Aminolevulinic Acid; Device: Blue light only
- Red Light only (Active Comparator): Red light only - no drug
  Interventions: Device: Red light only
- Blue light only (Active Comparator): Blue light only - no drug
  Interventions: Device: Blue light only

INTERVENTIONS:
Drug: 20 % Aminolevulinic Acid — topical medication for ALA-PDT and i-PDT
  Other Names: 5-Aminulevulinic acid HCl (ALA): Levulan® Kerastic® (Dusa Pharmaceuticals, Inc, Wilmington, MA, USA) (Dusa Pharmaceuticals)
  Arms: ALA-PDT; i-PDT
Device: Red light only — Red Light therapy
  Other Names: Omnilux Revive; 635 nm - LED (Phototherapeutics, Cheshire, UK)
  Arms: Red Light only
Device: Blue light only — Blue light only
  Other Names: Omnilux Blue; 415 nm LED (Phototherapeutics, Cheshire, UK)
  Arms: Blue light only; i-PDT

SUMMARY:
This research study aims to compare different methods for helping difficult to treat or scarring (cystic) acne, ALA-PDT and i-PDT.

There is an investigational procedure called photodynamic therapy (ALA-PDT) that has been reported to be very efficient for acne treatment since 2000. Photodynamic therapy (PDT) uses a drug called ALA (aminolevulinic acid), which is marketed as Levulan®.

Levulan® is applied directly to facial/back acne. This is the way that it is usually applied. Levulan® is left on the skin for three hours so the skin can absorb it. Next, the skin where the Levulan® was applied is exposed to a red light for activation.

The sebaceous glands get obstructed and inflamed causing acne. ALA gets down under your skin through the skin pores to where the glands are. PDT destroys the glands reducing the acne lesion.

Levulan® is absorbed by normal skin surrounding the oil glands. Therefore, this procedure also has some side effects. Some of the side effects include pain, burning sensation during the procedure, and redness, tenderness, and swelling after the procedure.

At Massachusetts General Hospital's Wellman Center for Photomedicine, the investigators developed another procedure called inhibitory-PDT (i-PDT) that is similar to ALA-PDT. i-PDT is aimed at reducing the side-effects of ALA- PDT.

The difference between these two procedures is that i-PDT uses a light source that will prevent Levulan® accumulation in the normal skin surface. The investigators would like to find out if Levulan® will be placed only inside the sebaceous glands.

DETAILED DESCRIPTION:
This is a pilot study to compare efficacy and side effects i-PDT and ALA-PDT. All subjects will receive ALA-PDT and i-PDT. Face or back regions will be divided into two sides, the right and left. One half of the face or back will receive ALA-PDT and the other half will receive i-PDT. For subjects with back acne, red light and blue light alone will be applied for comparison.

Healthy subjects with difficult to treat moderate or severe acne on the face or back are eligible to enroll.

The investigators will enroll about 35 patients at Massachusetts General Hospital (MGH) with follow-ups 1, 3 and 6 months after treatment.

ELIGIBILITY:
Inclusion criteria

1. Subjects with ages between 14 and 50 years, male or female.
2. Subjects with severe acne lesions (one or more nodules or cysts present) on their backs or face
3. Presence of moderate acne on the back and/or face that has been recalcitrant to previous treatments. Recalcitrant acne is acne with no or mild/temporary (less than 3 months) improvement after using:

   * Accutane® for at least one completed treatment cycle, and/or
   * Oral antibiotic for ≥ 3 months; and/or
   * Topical prescription retinoids (tretinoin - retinoic acid, adapalene, tazarotene or other derivatives) for ≥ 3 months, and/or
   * Topical benzoyl peroxide 2.5% or higher concentrations for ≥ 3 months
   * Hormonal treatments** for ≥ 3 months.
4. Willingness to participate in the study
5. Willingness to receive ALA-PDT treatment
6. Informed consent agreement signed by the subject
7. Willingness to follow the treatment schedule and post treatment care requirements
8. Willingness to not use topical or systemic (oral) anti-acne medications including medicated shampoo or soap during the study period.

Exclusion criteria

1. Subjects receiving concurrent oral retinoids or antibiotics

   ** Subjects with chronic use of antibiotics may be included if proven that its use has not changed the severity of their acne. AND

   *** Chronic use of antibiotic is considered ≥ 2 years of continuous use.
2. Scarring or infection of the area to be treated
3. Known photosensitivity
4. Presence of suntan in the area to be treated
5. Subjects who have taken medication known to induce photosensitivity in the previous 3 months
6. Subjects who have had prior oral retinoid (Accutane®) use within 6 months of entering the study
7. Prior oral antibiotic use within 1 month of entering the study (see exclusion #1)
8. Topical antibiotic or other topical anti-acne treatments use within 2 weeks of entering the study
9. Known anticoagulation or thromboembolic condition
10. Subjects who are immunosuppressed
11. Subject is unable to comply with treatment, home care or follow-up visits
12. Subject is pregnant or breast feeding
13. Subject has a history of being on photosensitive medications (thiazides [used to treat high blood pressure], tetracyclines, fluoroquinolones griseofulvin or sulfonamides [used to treat infections], sulfonylureas [used to treat diabetes], calcium channel blockers [used to treat hypertension]. phenothiazines [used to treat serious emotional problems]).
14. Known skin sensitivity to blue light
15. Porphyria (a disorder of the metabolism that can lead to sensitivity to light)
16. Allergies to chemicals called porphyrins
17. Subjects who started hormonal treatment (for medical conditions or birth control) within less than 3 months.

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2009-11-01 (Actual); Primary Completion 2013-09-01 (Actual); Study Completion 2014-12-01 (Actual)

PRIMARY OUTCOMES:
Efficacy: Investigator Global Assessment (IGA) scale for acne vulgaris | 0, 4, 8, 12, 16, 24 and 36 weeks
  0. Clear: No lesions but erythema and residual hyperpigmentation may be present
  1. Almost Clear: few scattered comedones and a few (< five) small papules
  2. Mild:< 50% face involved, many comedones/papules and pustules
  3. Moderate:> 50% of face involved. Numerous comedones, papules and pustules
  4. Severe: Entire face is covered with comedones, numerous papules and pustules and a few nodules and cysts.
  1) Clear or almost clear (Grades 0 or 1) as success at 12 weeks. 2) Two grade improvement as success at 12 weeks.

SECONDARY OUTCOMES:
Pain reduction | During, immediately after and 24 h after treatment
  Visual Pain Scale - 0 (no pain) -10 (severe pain)

OTHER OUTCOMES:
Side-effects Profile | Immediately after treatment and during follow-up visits
  Evaluation of overall side-effects of each test site